CLINICAL TRIAL: NCT07041827
Title: Cardiotoxicity and Other Late Effects After Radiotherapy and Immuno-chemoTherapy in Non-Hodgkin lYmphoma
Acronym: CLARITY
Status: Completed | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Other Study IDs: M18CNH; 10424 (Other Grant/Funding Number: KWF (Koningin Wilhelmina Fonds Kankerbestrijding))
Record Dates: First submitted 2019-02-20; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Non Hodgkin Lymphoma; DLBCL; Cardiovascular Diseases; Cardiomyopathies; Cardiotoxicity; Metabolic Syndrome; Quality of Life; Late Effect; Heart Failure
Keywords: Cardiotoxicity; Non-Hodgkin lymphoma; Late effects; Survivor
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Cardiovascular Diseases; Cardiomyopathies; Cardiotoxicity; Metabolic Syndrome; Heart Failure | interventions — Blood Specimen Collection; Echocardiography; Electrocardiography; Pulse Wave Analysis; Vascular Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — EDTA-plasma, serum, EDTA-whole blood (for DNA), citrate, heparin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Survivors: Over the past years, a Dutch multicentre hospital-based patient cohort of 5-year non-Hodgkin lymphoma survivors has been established. Survivors will be invited for the current study by their treating physician through the BETER survivorship clinics, or when patients have been dismissed from clinical follow-up, by their former treating physician (or head of the medical department, if the treating physician is retired) within each BETER clinic.
  Interventions: Diagnostic Test: Cardiovascular assessment
- Siblings: As there are no patients who are unexposed to potential cardiotoxic treatment in the BETER cohort we will request every participating NHL survivor to approach one of their siblings, more specifically the sibling who is closest in birthdate to the birthdate of the survivor, for participation in the study.
  Interventions: Diagnostic Test: Cardiovascular assessment

INTERVENTIONS:
Diagnostic Test: Cardiovascular assessment — A cardiovascular assessment will be performed to screen for (sub)clinical cardiovascular diseases and to compare the prevalences in survivors of non-Hodgkin lymphoma and a control group.
  Other Names: Blood & urine sampling (biomarkers); Echocardiography; Electrocardiography; Pulse wave velocity (arterial stiffness); EndoPAT (peripheral arterial tonometry - endothelial dysfunction); AGE-reader (advanced glycation end products); Questionnaires (cardiovascular risk factors & quality of life)

SUMMARY:
Survivors of non-Hodgkin lymphoma and a control group will be screened for (sub)clinical cardiovascular disease, to assess the influence of contemporary treatments on risk and burden of (sub)clinical cardiovascular disease and their influence on survival.

DETAILED DESCRIPTION:
Rationale: Few studies have thus far addressed the burden from treatment-related cardiovascular disease in long-term survivors of non-Hodgkin's lymphoma (NHL). The life expectancy of patients with aggressive B-cell NHL has significantly increased since treatment regimens have improved. Although the addition of rituximab to CHOP chemotherapy does not appear to increase cardiotoxicity during treatment, little is known about the long-term cardiac safety of R-CHOP. Nonetheless, cardiotoxicity due to doxorubicin exposure appears to be a key problem in clinical practice, while radiation exposure of the heart may add to cardiac disease risk.

Objective: The main objective is to assess in detail risk factors for cardiovascular disease and cardiotoxicity and to compare heart function parameters, vascular parameters and biomarkers associated with cardiovascular function among five- tot fifteen-year survivors, treated for aggressive B-cell NHL, and sibling controls and to assess the effects of cumulative doses of individual immuno- and chemotherapeutic agents and radiation of the heart on cardiovascular function parameters. Secondary objectives are to assess the prevalence of other late effects (metabolic syndrome, quality of life and the predictive value of newly developed markers for cardiovascular disease).

Study design: These parameters will be assessed in a cross-sectional study, nested in a well characterized cohort of aggressive B-cell NHL survivors, with a control population consisting of siblings of these survivors.

Study population: 350 survivors will be invited who are between five and fifteen years after treatment with (R-)CHOP with/without mediastinal radiotherapy, and compare them with 175 sibling controls. Eligible participants will be approached and invited to the BETER clinic by their (former) treating physician.

Main study parameters/endpoints: The main study parameters will be echocardiographic systolic and diastolic heart parameters and global longitudinal strain measurement, arterial stiffness (by pulse wave velocity measurements), endothelial function (by peripheral arterial tonometry), electrocardiography, advanced glycation end products (by skin autofluorescence, AGE-reader), presence of (sub)clinical cardiovascular disease and biomarkers. Adverse cardiovascular events, risk factors and quality of life will be assessed through questionnaires and physical measurements. Exposure to (R-)CHOP and radiotherapy will be extracted from the medical history. Multivariable logistic and linear regression analyses will be used for analyses.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: With the results of our study, guidelines for follow up and prevention will be developed which will benefit the participants during their own follow up in the future. The burden of participating is expected to be low since the study is mainly observational and assessments required in the context of research as much as possible combined with the provided standard of care for survivors during one or two hospital visits.

ELIGIBILITY:
Inclusion Criteria (survivors):

* 5-15 year survivors from the patient cohort with (mediastinal) large B-cell non-Hodgkin lymphoma (ICD-code 9679) or diffuse large B-cell non-Hodgkin lymphoma (ICD-code 9684), treated with R-CHOP:

  * 200 survivors treated between five to ten years ago (2007-2012)
  * 150 survivors treated between ten to fifteen years ago (2002-2007)
* Treated in one of the following centers: AVL, Amsterdam UMC (location VUmc or AMC), LUMC, EMC, UMCU, UMCG, UMC Radboud.
* Age at diagnosis 15 up to 60 years.
* Age at the time of inclusion: younger than 75 years old.

Exclusion criteria (survivors):

* Use of immunosuppressant and/or prednisolone
* HIV-infected individuals
* Pregnant women
* Mental disability or psychological condition potentially hampering compliance with the study protocol
* Insufficient understanding of the Dutch language

Inclusion criteria (siblings):

175 siblings of the above mentioned patients (maximum of 1 sibling per patient) with their date of birth closest to the birthdate of the survivor.

Exclusion Criteria (siblings):

* Use of immunosuppressant and/or prednisolone
* HIV-infected individuals
* Pregnant women
* Mental disability or psychological condition potentially hampering compliance with the study protocol
* Insufficient understanding of the Dutch language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Survivors: Over the past years, a Dutch multicentre hospital-based patient cohort of 5-year non-Hodgkin lymphoma survivors has been established. Survivors will be invited for the current study by their treating physician through the BETER survivorship clinics, or when patients have been dismissed from clinical follow-up, by their former treating physician (or head of the medical department, if the treating physician is retired) within each BETER clinic.
  * Siblings: As there are no patients who are unexposed to potential cardiotoxic treatment in the BETER cohort we will request every participating NHL survivor to approach one of their siblings, more specifically the sibling who is closest in birthdate to the birthdate of the survivor, for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Echocardiography: systolic and diastolic heart parameters, various strain measurements such as global longitudinal strain | Once, at enrollment
  LVEF (continuous), LVEF<50%, GLS (continuous) GLS>-18%, NT-proBNP (continuous), NT-proBNP>=125 pg/mL

SECONDARY OUTCOMES:
Electrocardiography | Once, at enrollment
  Presence of cardiac disease
Pulse wave velocity | Once, at enrollment
  Measurement of arterial stiffness / vascular function
Association of different biomarkers | Once, at enrollment
  Value of different biomarkers (Nt-proBNP, Troponin T, sST2, galectin-3, GDF-15, high sensitive CRP)
EndoPAT (peripheral arterial tonometry) | Once, at enrollment
  Measurement of endothelial function / vascular function
Metabolic syndrome | Once, at enrollment
  Defined if 3 out of 5 of the following criteria are present: hypertension, dyslipidemia, diabetes, obesity, increased abdominal circumference
Questionnaires | Once, at enrollment
  Assessment of health related quality of life and symptoms by validated questionnaires: EORTC QLQ-C30, EORTC-NHL-HG29, EORTC-BR29/PR-25 (sexuality items)
Advanced glycation end products | Once, at enrollment
  Assessment of AGEs by skin autofluorescence, as a marker for cardiovascular and metabolic disease

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schaapveld, PhD, Study Director — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided